CLINICAL TRIAL: NCT02355886
Title: Randomized Placebo Control Trial of Perioperative Gabapentin to Reduce Total Analgesic Requirements in Patients Undergoing Radical Cystectomy
Brief Title: Gabapentin in Reducing the Need for Pain Medication in Patients With Bladder Cancer Undergoing Radical Cystectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 9274; NCI-2015-00083 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9274 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Results first posted 2019-06-04 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Bladder Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (gabapentin) (Experimental): Patients receive gabapentin PO TID for 48 hours after surgery.
  Interventions: Drug: Gabapentin; Other: Questionnaire Administration
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO TID for 48 hours after surgery.
  Interventions: Other: Placebo; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Gabapentin — Given PO
  Other Names: Gralise; Neurontin
  Arms: Arm I (gabapentin)
Other: Placebo — Given PO
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II/III trial studies gabapentin in reducing the need for pain medication in patients with bladder cancer undergoing surgery to remove the bladder and nearby tissue and organs. Gabapentin may reduce the amount of pain medicine required after surgery, improve pain after surgery, and/or reduce the length of hospital stay after surgery.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess if perioperative gabapentin will decrease post-operative analgesic requirements within the first 48 hours after radical cystectomy (RC) in patients undergoing RC as measured morphine equivalents.

SECONDARY OBJECTIVES:

I. To assess patient self-assessment of postoperative pain on Numeric Pain Scale (NPS) at 24 and 48 hours.

II. To assess time to return of bowel function (ROBF).

III. To assess length of stay (LOS) following RC.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive gabapentin orally (PO) thrice daily (TID) for 48 hours after surgery.

ARM II: Patients receive placebo PO TID for 48 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bladder cancer
* Anticipated radical cystectomy with ileal conduit or orthotopic neobladder

Exclusion Criteria:

* Presence of spinal cord injury including any form of paraplegia or quadriplegia
* Allergy to gabapentin
* Active alcohol dependence, defined as 2 or more positive questions on the CAGE alcoholism questionnaire
* Illicit drug use (excluding recreational marijuana)
* Chronic kidney disease with glomerular filtration rate < 30 ml/min
* Pregnancy: All female patients < 55 years old (yo) will be administered a urine pregnancy test prior to enrollment
* Non-English speaking patients
* Chronic gabapentin, or the similar drug pregabalin, use
* Chronic narcotic use (daily or near daily use for > 90 days)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-04-22 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2019-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Wright, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Gabapentin) | Arm II (Placebo)
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Gabapentin) | Arm II (Placebo) | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.82 (9.69) | 68.33 (8.39) | 67.5 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 12 | 6 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 12 | 25
  More than one race | 00 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25
neoadjuvant chemotherapy [Count of Participants; unit: Participants] | 2 | 6 | 8

OUTCOME MEASURES:

1. Primary Outcome: Patient Total Equivalent Analgesic Requirement (Morphine Equivalents)
Description: Geometric Mean and Standard Deviation of patient total equivalent analgesic
Time Frame: 48 hours post-radical cystectomy
Measure: Geometric Mean (Standard Deviation); unit: Total oral morphine equivalents in mg
Arm/Group | Arm I (Gabapentin) | Arm II (Placebo)
Number analyzed (Participants) | 13 | 12
Total oral morphine equivalents in mg | 297.65 (179.95) | 396.16 (149.84)

2. Secondary Outcome: Length of Stay Following Radical Cystectomy
Description: The two study groups will be compared by Length of stay following radical cystectomy
Time Frame: duration of hospital stay. Days to weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm I (Gabapentin) | Arm II (Placebo)
Number analyzed (Participants) | 13 | 12
days | 6.58 (1.98) | 6.73 (2.83)

3. Secondary Outcome: Patient Self-assessed Pain on Numerical Pain Scale
Description: The two study groups compared on Patient self-assessed pain on numerical pain likert scale. Numeric Pain Scale was utilized with values of 0-10 with increasing severity.
Time Frame: Up to 48 hours post-radical cystectomy
Measure: Mean (Standard Deviation); unit: Sore on a scale
Arm/Group | Arm I (Gabapentin) | Arm II (Placebo)
Number analyzed (Participants) | 13 | 12
Sore on a scale | 5.15 (2.8) | 7.67 (1.89)

ADVERSE EVENTS:
Time Frame: an average of one week
Arm/Group | Arm I (Gabapentin) | Arm II (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 6/13 | 10/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Gabapentin) (N=13) | Arm II (Placebo) (N=12)
nausea (Gastrointestinal disorders) | 3 (3) | 10 (10)
sedation (Nervous system disorders) | 5 (5) | 1 (1) — PACU sedation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-20): https://cdn.clinicaltrials.gov/large-docs/86/NCT02355886/Prot_SAP_000.pdf